CLINICAL TRIAL: NCT06105567
Title: The Effect of Education Given According to the Health Promotion Model on Premenstrual Symptoms, Emotional Eating Behavior and Perceived Stress
Acronym: Premenstrual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Cansu Mine Aydin, research assistant, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KAFKAS-SAG-CMAYDIN-002
Record Dates: First submitted 2023-10-16; First posted 2023-10-27 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Premenstrual Syndrome; Emotional Disorder; Perceived Stress
Keywords: premenstrual syndrome; emotional eating; health promotion model
MeSH Terms: conditions — Premenstrual Syndrome; Emotional Eating | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The research will be conducted as a pretest-posttest randomized controlled study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Effect of Education on Premenstrual Symptoms, Emotional Eating Behavior and Perceived Stress (Experimental): Students who score over 110 on the premenstrual syndrome scale and meet the study criteria will be included in the experimental and control groups. Personal Information Form, PMS Scale, Premenstrual Eating Habits Form, Healthy Lifestyle Behaviors Scale, Emotional Eating Scale, Perceived Stress Scale and Visual Visual Pain Scale will be administered to the students in this group before the training. Premenstrual syndrome periods will be determined by creating a menstrual cycle calendar for the participants. Students will be trained with their first powerpoint presentation. Afterwards, brochures will be distributed. It will be applied according to the Philips 66 technique. 4 weeks after the first training, students will be given general reminder training online during pms periods. Survey forms will be filled out by the group 4 weeks after the second training.
  Interventions: Behavioral: Training given according to the health promotion model by applying the Philips 66 technique
- control group (No Intervention): Students who score over 110 on the premenstrual syndrome scale and meet the study criteria will be included in the experimental and control groups. Students in this group will not receive training and will be administered the Personal Information Form, PMS Scale, Premenstrual Eating Habits Form, Healthy Lifestyle Behaviors Scale, Emotional Eating Scale, Perceived Stress Scale and Visual Vissual Pain Scale. Data will be collected by face-to-face research method. Survey forms will be filled out by the control group.

INTERVENTIONS:
Behavioral: Training given according to the health promotion model by applying the Philips 66 technique — The Effect of Education Given According to the Health Promotion Model on Premenstrual Symptoms, Emotional Eating Behavior and Perceived Stress
  Other Names: control group; health promotion model; Philips 66 technique
  Arms: Effect of Education on Premenstrual Symptoms, Emotional Eating Behavior and Perceived Stress

SUMMARY:
Nurses have important duties in this regard due to their roles such as health education, health protection, development and consultancy.

In this study, it is thought that the training given according to the health promotion model will both create a resource for nurses and contribute to the literature with the results obtained by applying this training to people experiencing PMS.The research will be conducted as a pretest-posttest randomized controlled study.

H1: Education given according to the health promotion model has an effect on premenstrual symptoms, emotional eating behavior and perceived stress.

H0: Education given according to the health promotion model has no effect on premenstrual symptoms, emotional eating behavior and perceived stress.

The total number of students in the research population is 330.In the G*Power 3.1.9.7 program, for the effect size t test, d = 0.94, alpha (α) = 0.05, and power (1-β) = 0.95, and the minimum total sample number was determined as 52, experimental group: 26, control group: 26. . However, taking into account the losses in the study, a total of 60 people will be included in the study. (experiment:30, control:30).

The first group will be divided into the group trained according to the health promotion model using the Philips 66 technique, and the second group will be divided into the control group.

DETAILED DESCRIPTION:
Changes that gradually disappear with the onset of menstruation in women are called premenstrual syndrome.In this syndrome, anxiety, irritability, lack of concentration, depression, mood swings, drowsiness, sleep disturbance, breast tenderness, appetite change, bloating, headache, weight gain, abdominal pain, fatigue and gastrointestinal symptoms are observed. Since these symptoms negatively affect both the work and personal lives of women, safe and effective treatments are needed. In this case, many women report using exercise as a strategy to help them cope with PMS, and exercise is often recommended for symptom management.PMS can also play a role in symptoms by affecting the individual's food choices. Emotional eating behavior is defined as a person's use of food as an escape from negative emotions and can lead to many conditions such as obesity, eating disorders and hormonal problems. Health promotion means increasing one's control over one's health by improving one's own health. It enables the individual to improve their physical and social environment, change their behavior, and reach the best level of physical and mental health. Philips 66 technique is a process based on active learning, problem and collaborative learning theory, student-centered, and uses the best learning techniques to improve students' performance and realize meaningful learning activity. It is among the responsibilities of healthcare personnel to identify the factors that negatively affect women's lives in order to ensure continuity of health, ease of premenstrual symptoms, and to use the findings to improve women's health. Nurses have important duties in this regard due to their roles such as health education, health protection, development and consultancy. In this study, it is thought that the training given according to the health promotion model will both create a resource for nurses and contribute to the literature with the results obtained by applying this training to people experiencing PMS.Nurses have important duties in this regard due to their roles such as health education, health protection, development and consultancy.In this study, it is thought that the training given according to the health promotion model will both create a resource for nurses and contribute to the literature with the results obtained by applying this training to people experiencing PMS.The research will be conducted as a pretest-posttest randomized controlled study.

H1: Education given according to the health promotion model has an effect on premenstrual symptoms, emotional eating behavior and perceived stress.

H0: Education given according to the health promotion model has no effect on premenstrual symptoms, emotional eating behavior and perceived stress.

The total number of students in the research population is 330.In the G*Power 3.1.9.7 program, for the effect size t test, d = 0.94, alpha (α) = 0.05, and power (1-β) = 0.95, and the minimum total sample number was determined as 52, experimental group: 26, control group: 26. . However, taking into account the losses in the study, a total of 60 people will be included in the study. (experiment:30, control:30).

The first group will be divided into the group trained according to the health promotion model using the Philips 66 technique, and the second group will be divided into the control group.In the first stage, the "Premenstrual Syndrome Scale" will be applied to the students and the students will be placed in the experimental and control groups. In the second stage, Personal Information Form, PMS Scale, Premenstrual Eating Habits Form, Healthy Lifestyle Behaviors Scale, Emotional Eating Scale, Perceived Stress Scale and Visual Vissual Pain Scale will be applied to the students in this group before training. Data will be collected by face-to-face research method. Premenstrual syndrome periods will be determined by creating a menstrual cycle calendar for the participants. In the third stage, students in the experimental group will be trained with the first powerpoint presentation. Then brochures will be distributed. It will be applied according to the Philips 66 technique. In the fourth stage, 4 weeks after the first training, general reminder training will be given online during students' pms periods. In the fifth stage, 4 weeks after the second training, survey forms will be filled out by the experimental group and the control group.

ELIGIBILITY:
Inclusion Criteria:

Getting over 110 points from the PMS scale,

* Experiencing at least five PMS symptoms every month,
* Not having had sexual intercourse
* Regular menstruation, (regular menstruation (between 21-35 days))
* Not having any chronic disease,
* Not using any method to cope with PMS
* Not taking Hormone Replacement Therapy
* Women who agreed to participate in the study were included in the study group.

Exclusion Criteria:

* • Having had sexual intercourse,

  * Allergy,
  * Irregular menstruation,
  * Not having regular menstrual periods in the last three months,
  * Having received a psychiatric diagnosis,
  * Do not have any gynecological disease (abnormal uterine bleeding, myoma, ovarian cyst, etc.)
  * Using contraceptive medication,
  * 1st and 4th year nursing and midwifery students

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — premenstrual syndrome
Enrollment: 86 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale (PMSS) | 3 month
  Participants in the study will be asked to fill out this scale in the 1st and 8th weeks. Women with premenstrual syndrome will be included in the study. The total score is obtained from the sum of the scores from all sub-dimensions. A minimum of 44 points and a maximum of 220 points can be obtained from the scale. An increase in the score obtained from the scale indicates that the intensity of the symptoms increases. PMS is considered "present" if the total scale score (220) on the PMS scale exceeds 50% (110).
Eating Habits During the Premenstrual Period Form | 3 month
  The form created by the researchers covering the change in food consumption during the PMS period consists of a total of 15 questions.Since there is no scale, there is no low or high score.
Healthy Lifestyle Behaviors Scale | 3 month
  The scale, which determines people's health-improving behaviors regarding their healthy lifestyle, consists of 48 items and 6 subgroups. The lowest total score of the scale, which has all positive items and 4 answer options, is 48 and the highest total score is 192.
Emotional Eating Scale | 3 month
  Emotional eating is defined as a coping strategy with negative emotions and experiences.The lowest score that can be obtained from the single-factor scale is 14 and the highest score is 70.
  Individuals who score 35 points and above from the scale are considered to have emotional eating.
Perceived Stress Scale | 3 month
  It shows how stressful the individual perceives the events he encounters.Scoring of the scale varies between 0 and 56, with a high score indicating that the individual has a high perception of stress.
Visual comparison scale | 3 month
  They were asked to question the existence of pain and to mark it on this scale by explaining the pain expressed by the points on it.The lowest score is 1 and the highest is 10, and as the score increases, the pain level increases.
Personal Information Form | 3 month
  The form prepared by the researchers consists of 3 sections and 46 questions.

SECONDARY OUTCOMES:
Feedback of the training using the Health Promotion Model and Philips 66 technique | 1 year
  It will be filled out by the participants at the end of the training in the 8th week.
Eating Habits During the Premenstrual Period Form | 1 year
  The form will be filled out again in the 4th and 8th weeks of the study.The form created by the researchers covering the change in food consumption during the PMS period consists of a total of 15 questions.Since there is no scale, there is no low or high score.
Premenstrual Syndrome Scale (PMSS) | 1 year
  Participants in the study will be asked to fill out this scale in the 8th weeks. Women with premenstrual syndrome will be included in the study. The total score is obtained from the sum of the scores from all sub-dimensions. A minimum of 44 points and a maximum of 220 points can be obtained from the scale. An increase in the score obtained from the scale indicates that the intensity of the symptoms increases. PMS is considered "present" if the total scale score (220) on the PMS scale exceeds 50% (110).
Healthy Lifestyle Behaviors Scale | 1 year
  The scale will be applied at the 8th week. The scale, which determines people's health-improving behaviors regarding their healthy lifestyle, consists of 48 items and 6 subgroups. The lowest total score of the scale, which has all positive items and 4 answer options, is 48 and the highest total score is 192.
Emotional Eating Scale | 1 year
  The scale will be applied at the 8th week.Emotional eating is defined as a coping strategy with negative emotions and experiences.The lowest score that can be obtained from the single-factor scale is 14 and the highest score is 70. Individuals who score 35 points and above from the scale are considered to have emotional eating.
Perceived Stress Scale | 1 year
  The scale will be applied at the 8th week.It shows how stressful the individual perceives the events he encounters.Scoring of the scale varies between 0 and 56, with a high score indicating that the individual has a high perception of stress.
Visual comparison scale | 1 year
  The scale will be applied at the 8th week.They were asked to question the existence of pain and to mark it on this scale by explaining the pain expressed by the points on it.The lowest score is 1 and the highest is 10, and as the score increases, the pain level increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafkas University, Kars, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No